CLINICAL TRIAL: NCT01301339
Title: A1c FIT TEST: An Epidemiological Study Correlating Hemoglobin A1c With Results of the Air Force Physical FITness TEST.
Status: Completed | Type: Observational
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FWH20110007H
Record Dates: First submitted 2011-02-17; First posted 2011-02-23 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Pre-Diabetes; Diabetes; Cardiovascular Risks
Keywords: Pre-Diabetes; Diabetes; cardiovascular risks
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- failed and passed physical fitness test: 520 subjects who have failed their Air Force physical fitness test and 520 volunteers who have passed their physical fitness test both within the last 6 months

SUMMARY:
The purpose of this study is to evaluate the prevalence of pre-diabetes and diabetes among those Air Force personnel who have not passed the Air Force physical fitness test (AFPT) and to evaluate the usefulness of the AFPT as a prescreening tool for these disease processes.

ELIGIBILITY:
Inclusion:

* Tricare Insurance Beneficiary (military insurance) receiving care at Nellis AFB
* Over the age of 18 and took their AFPT within the past 1 month.

Exclusion:

* Previous diagnosis of diabetes
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Active duty Air Force personnel will be recruited from all male and female patients 18 years or older at the Mike O'Callaghan Federal Hospital. A total of 1040 subjects will be recruited (520 subjects who have failed their Air Force physical fitness test and 520 volunteers who have passed their physical fitness test both within the last 6 months from recruitment into this study).
Sampling Method: Non-Probability Sample
Enrollment: 535 (Actual)
Dates: Start 2011-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Do Air Force personnel who fail the Air Force physical fitness test have a higher incidence of pre-diabetes than those who pass the test? | within 1 year
  Do Air Force personnel who fail the Air Force physical fitness test have a higher incidence of pre-diabetes than those who pass the test?

SECONDARY OUTCOMES:
And for those who fail, do they have higher cardiovascular risks as correlated with fasting lipid panel. | within 1 year
  And for those who fail, do they have higher cardiovascular risks as correlated with fasting lipid panel.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Timboe, D.O., Principal Investigator — Mike O'Callaghan Federal Hospital/Nellis Air Force Base
Locations (1):
- Mike O'Callaghan Federal Hospital/Nellis Air Force Base, Las Vegas, Nevada, United States